CLINICAL TRIAL: NCT03845465
Title: Positive Psychology Intervention to Treat Diabetes Distress in Teens With Type 1 Diabetes
Acronym: T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190020
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Active Comparator): Participants in the Education group will complete a behavioral health contract and will receive an educational packet.
  Interventions: Behavioral: Education
- PA + Education (Experimental): Participants in the Positive Affect + Education group will complete a behavioral health contract and receive an educational packet. In addition, they will receive intervention components aimed at inducing positive affect.
  Interventions: Behavioral: Positive Affect + Education; Behavioral: Education

INTERVENTIONS:
Behavioral: Positive Affect + Education — Adolescents will complete a health behavior contract and receive an educational packet at baseline. Adolescents will complete a positive affect interview at baseline. They will receive automated text messages 5 days/week for 8 weeks. Messages will be tailored to include adolescents' responses to the baseline interview, including reminders to engage in gratitude and self-affirmation. Additionally, to induce positive mood they will be texted gift cards codes valued at $5.00. Further, caregivers will be asked to provide weekly positive affirmations to their adolescents, focused on non-diabetes strengths.
  Arms: PA + Education
Behavioral: Education — Adolescents will complete a health behavior contract and receive an educational packet with information about diabetes management.

SUMMARY:
The treatment regimen for type 1 diabetes is complex and demanding, and many adolescents experience diabetes distress related to the daily demands of diabetes care, which can cause problems with diabetes management and glycemic control. The proposed study will conduct a multisite, randomized trial to test the effects of a positive psychology intervention aimed at treating diabetes distress and improving glycemic outcomes. The potential benefits include helping adolescents achieve better glycemic control, improved self-management, and psychosocial outcomes

DETAILED DESCRIPTION:
Adolescents with type 1 diabetes (T1D) struggle to meet treatment goals - only 17% met the target for glycemic control in a recent national study - and many adolescents experience high levels of diabetes distress related to the daily demands of diabetes care. Yet, previous interventions to improve glycemic control in adolescents with type 1 diabetes have only shown modest to moderate effects, and many have been time-intensive and expensive. Thus, there is a need for novel interventions to improve outcomes in adolescents with T1D. Increasing positive affect, or pleasurable engagement with the environment (e.g., feeling happy, cheerful, proud), has been shown to promote the use of more adaptive coping strategies to manage stress. Thus, the proposed study is based on the premise that, by boosting positive affect in teens with diabetes, we will enhance the use of adaptive coping strategies and reduce diabetes distress, thereby improving glycemic control in adolescents. Through an iterative series of pilot studies, our research team adapted a behavioral intervention using a positive psychology framework that we demonstrated to be feasible and acceptable for adolescents with T1D. This intervention is aimed at inducing positive affect in adolescents (age 13-17) through empirically-validated, tailored exercises in gratitude, self-affirmation, and caregiver affirmations. In our pilot studies, the intervention had promising effects on adolescents' quality of life, diabetes-related stress, and family conflict, all of which are closely linked with diabetes distress. We now plan to evaluate the efficacy of the intervention in a multisite, randomized controlled trial. The aims of this study are to 1) evaluate the effects of a positive psychology intervention for adolescents (age 13-17) and their caregivers on glycemic control; 2) evaluate the effects of the intervention on diabetes distress, coping, and self-care behavior; and 3) explore the differential impact of intervention effects across demographic and treatment variables. We plan to randomize 200 adolescent-caregiver dyads to the Positive Affect + Education intervention (n=100) or the Education only intervention (n=100) from two clinical sites (Vanderbilt University Medical Center and Children's National Medical Center). By employing a positive psychology framework, we propose an innovative approach to treat diabetes distress and improve glycemic outcomes. We believe this novel intervention has the potential to improve outcomes in adolescents with T1D, and the use of automated text messaging to deliver the intervention offers possibilities for wide dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17
* Diagnosed with type 1 diabetes for at least 12 months
* Speak and read English
* Report at least moderate diabetes distress on the Problem Areas in Diabetes Scale - Teen version

Exclusion Criteria:

- Other serious health conditions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's National, Washington D.C., District of Columbia
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straton E, Anifowoshe K, Moore H, Streisand R, Jaser SS. Associations of Coping Strategies With Glycemic and Psychosocial Outcomes Among Adolescents With Type 1 Diabetes Experiencing Diabetes Distress. Ann Behav Med. 2024 Aug 7;58(9):628-633. doi: 10.1093/abm/kaae028. PMID 39014980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from pediatric diabetes clinics at Vanderbilt University Medical Center and Children's National Hospital.
Pre-assignment Details: Caregiver-adolescent dyads were enrolled and randomized. Protocol Enrollment, Number Started, and Completed reflect participants.
  Two dyads were enrolled but not randomized:
  * One caregiver-adolescent dyad gave informed consent but did not finish baseline data and did not respond to the study team.
  * One caregiver-adolescent dyad gave informed consent and completed baseline data but were found to be ineligible because the teen did not have access to a cell phone.
Period: Baseline Through Intervention
Arm/Group | Education | PA + Education
Started (400 individuals were enrolled, but only 396 were randomized. 2 individuals gave informed consent but did not finish baseline data. 2 individuals gave informed consent and completed baseline data but were found to be ineligible.) | 198 | 198
Caregivers | 99 | 99
Adolescents | 99 | 99
Completed | 194 | 198
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0
Period: 3-month Data Collection
Arm/Group | Education | PA + Education
Started | 194 | 198
Caregivers | 97 | 99
Adolescents | 97 | 99
Completed | 194 | 198
Not Completed | 0 | 0
Period: 6-month Data Collection
Arm/Group | Education | PA + Education
Started | 194 | 198
Caregivers | 97 | 99
Adolescents | 97 | 99
Completed | 194 | 196
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: 12-month Data Collection
Arm/Group | Education | PA + Education
Started | 194 | 196
Caregivers | 97 | 98
Adolescents | 97 | 98
Completed | 194 | 194
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants were caregiver-adolescent dyads.
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | PA + Education | Total
Number analyzed (Participants) | 198 | 198 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Caregiver age analyzed separately from adolescent age.
  years
    Adolescent Age: number analyzed (Participants) | 99 | 99 | 198
    Adolescent Age | 15.4 (1.4) | 15.3 (1.4) | 15.3 (1.4)
    Caregiver Age: number analyzed (Participants) | 99 | 99 | 198
    Caregiver Age | 46.1 (7.1) | 45.3 (7.6) | 45.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Caregiver sex analyzed separately from adolescent sex. 1 caregiver did not report sex.
  Participants
    Adolescent Sex: number analyzed (Participants) | 99 | 99 | 198
    Adolescent Sex: Female | 57 | 58 | 115
    Adolescent Sex: Male | 42 | 41 | 83
    Caregiver Sex: number analyzed (Participants) | 98 | 99 | 197
    Caregiver Sex: Female | 84 | 85 | 169
    Caregiver Sex: Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregiver ethnicity analyzed separately from adolescent ethnicity.
  Participants
    Adolescent Ethnicity: number analyzed (Participants) | 99 | 99 | 198
    Adolescent Ethnicity: Hispanic or Latino | 7 | 2 | 9
    Adolescent Ethnicity: Not Hispanic or Latino | 92 | 97 | 189
    Adolescent Ethnicity: Unknown or Not Reported | 0 | 0 | 0
    Caregiver Ethnicity: number analyzed (Participants) | 99 | 99 | 198
    Caregiver Ethnicity: Hispanic or Latino | 5 | 2 | 7
    Caregiver Ethnicity: Not Hispanic or Latino | 93 | 95 | 188
    Caregiver Ethnicity: Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregiver race analyzed separately from adolescent race.
  Participants
    Adolescent Race: number analyzed (Participants) | 99 | 99 | 198
    Adolescent Race: American Indian or Alaska Native | 1 | 1 | 2
    Adolescent Race: Asian | 3 | 5 | 8
    Adolescent Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescent Race: Black or African American | 23 | 24 | 47
    Adolescent Race: White | 63 | 60 | 123
    Adolescent Race: More than one race | 8 | 8 | 16
    Adolescent Race: Unknown or Not Reported | 1 | 1 | 2
    Caregiver Race: number analyzed (Participants) | 99 | 99 | 198
    Caregiver Race: American Indian or Alaska Native | 1 | 1 | 2
    Caregiver Race: Asian | 3 | 6 | 9
    Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Caregiver Race: Black or African American | 21 | 20 | 41
    Caregiver Race: White | 70 | 67 | 137
    Caregiver Race: More than one race | 2 | 3 | 5
    Caregiver Race: Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — Caregiver Region of Enrollment Population: Caregiver region of enrollment.
  participants
    United States: number analyzed (Participants) | 99 | 99 | 198
    United States | 99 | 99 | 198
Region of Enrollment [Number; unit: participants] — Adolescent region of enrollment Population: Adolescent region of enrollment
  participants
    United States: number analyzed (Participants) | 99 | 99 | 198
    United States | 99 | 99 | 198
Diabetes Distress (PAID-T) [Mean (Standard Deviation); unit: score on a scale] — Problem Area in Diabetes - Teen (PAID-T) consists of 14 items measuring adolescents' diabetes distress. Scores range from 14-84, and higher scores indicate greater distress. A score of 44 or higher indicates clinically significant distress. Population: Diabetes distress was collected from adolescent participants (not caregivers).
  score on a scale
    number analyzed (Participants) | 99 | 99 | 198
    (all) | 48.4 (10.3) | 48.3 (10.7) | 48.4 (10.5)
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — Hemoglobin A1c measured as part of clinic visit indicates the amount of glucose attached to hemoglobin. Population: HbA1c values not available for all adolescent participants due to COVID-related disruptions to clinical care.
  percentage of glycated hemoglobin
    number analyzed (Participants) | 93 | 94 | 187
    (all) | 9.4 (2.0) | 8.9 (2.3) | 9.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c measures the amount of glucose attached to hemoglobin. It is assessed as part of regular diabetes clinic visits. The target is <7.0%.
Time Frame: 3 months
Population: A1c only collected from adolescents participants (not caregivers), since adolescents had type 1 diabetes. A1c was not available for all participants, due to COVID-related disruptions to diabetes clinic visits.
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 85 | 89
Percentage of glycated hemoglobin | 9.0 (2.0) | 9.0 (2.4)

2. Secondary Outcome: Diabetes Distress
Description: The Problem Area In Diabetes - Teen (PAID-T) measures diabetes distress. Scores range from 14-84, with higher scores indicated greater distress. A total score of 44 or higher is considered clinically significant.
Time Frame: 3 months
Population: Only adolescent participants completed this measure. Data were not collected from all participants at the 3-month time point due to COVID-related disruptions to diabetes clinic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
score on a scale | 43 (16) | 45 (14)

3. Secondary Outcome: Primary Control Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher scores indicate greater relative use of primary control coping (e.g., problem solving, emotional modulation).
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ratio score
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
ratio score | .16 [.14 to .18] | .16 [.13 to .18]

4. Secondary Outcome: Secondary Control Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of secondary control coping (e.g., acceptance, distraction, positive thinking).
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ratio score
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
ratio score | .24 [.20 to .27] | .23 [.21 to .26]

5. Secondary Outcome: Disengagement Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of disengagement coping (e.g., avoidance, denial).
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ratio score
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
ratio score | .16 [.14 to .17] | .16 [.14 to .18]

6. Secondary Outcome: Positive Affect
Description: Positive affect measured using the Positive and Negative Affect Scale for children (PANAS-C). The positive affect scale consists of 15 items, which are summed for a total score, ranging from 15-60. Higher scores indicate higher levels of positive affect.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
score on a scale | 41 (11) | 44 (11)

7. Secondary Outcome: Diabetes Self-Care Behavior
Description: The Self Care Inventory measures adherence to the recommended diabetes treatment regimen. Adolescents and parents report on the adolescents' self-care behaviors. A mean score is calcuated, ranging from 1-5. Higher scores indicate higher levels of self-management behaviors.
Time Frame: 3 months
Population: Data were not collected from all participants at the 3-month time point due to COVID-related disruptions to diabetes clinic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
score on a scale | 3.74 (0.65) | 3.72 (0.68)

8. Secondary Outcome: Diabetes-Related Quality of Life
Description: Type 1 Diabetes and Life measures adolescents self-reported diabetes-related quality of life. Scores range from 0-100, and higher scores indicate better quality of life.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education | PA + Education
Number analyzed (Participants) | 91 | 87
score on a scale | 52 (14) | 52 (14)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the active study period (4 years).
Description: Adverse events were self-reported by adolescent participants. We did not collect adverse events from caregivers.
Arm/Group | Education | PA + Education
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 0/99 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT03845465/Prot_SAP_000.pdf